CLINICAL TRIAL: NCT02846558
Title: A Pragmatic Trial of Dietary Programs in People With Multiple Sclerosis
Brief Title: A Pragmatic Trial of Dietary Programs in People With Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00105123
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Multiple Sclerosis
Keywords: calorie restriction; weight loss
MeSH Terms: conditions — Multiple Sclerosis; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Calorie Restriction - Frequent Patient Communication (Experimental): MS patients receiving monthly natalizumab infusions will use the LoseIt! smartphone application to log daily food consumption. Data from the app will be collected at follow-up visits. Patients will receive initial training in using the app, and then receive weekly supportive messages encouraging them to adhere to the calorie restriction diet between 3- and 6-month followup visits. Results will be compared primarily to those collected from the Standard of Care arm.
  Interventions: Other: Frequent Patient Interaction; Device: LoseIt! Smartphone Application
- Timing Restriction (Experimental): MS patients receiving monthly natalizumab infusions who are ineligible for the calorie restriction portion of the study (the Frequent Patient Activation and Standard of Care arms) will be offered the option to enroll in the second part of the study, assessing differences in outcomes between daily 16-hour fasting periods and no dietary changes. Patients in the second part of the study randomized to this arm will consume their normal daily food intake, but restrict eating to an 8-hour period during the day. Results will be compared to patients who do not make any changes to their diet, the No Change arm.
  Interventions: Behavioral: Timing Restriction
- Calorie Restriction - Communication Standard of Care (Placebo Comparator): MS patients receiving monthly natalizumab infusions will use the LoseIt! smartphone application to log daily food consumption. Data from the app will be collected at follow-up visits. Besides initial training with the application and 3- and 6-month follow up exams, participants will not receive additional support or interaction from the study team.Results will be compared with those collected from the Frequent Patient Interaction arm.
  Interventions: Device: LoseIt! Smartphone Application
- No Diet Change (No Intervention): MS patients receiving natalizumab infusions who were ineligible for the calorie restriction portion of the study (e.g. body mass index < 25 kg/m^2) or did not wish to participate in calorie restriction, may elect to be part of the second portion of the study. If so, they may be randomized to this arm, in which no changes are made to amount or timing of daily food intake. Results will be compared with the experimental Timing arm

INTERVENTIONS:
Other: Frequent Patient Interaction — Weekly informational and supportive text messages will be sent to patients, encouraging adherence to the calorie restriction diet.
  Arms: Calorie Restriction - Frequent Patient Communication
Behavioral: Timing Restriction — Patients continue to follow their normal diet, but limit food intake to an 8-hour period during the day.
  Arms: Timing Restriction
Device: LoseIt! Smartphone Application — Patients will be trained by study staff to download the LoseIt! application, and use it to log all food intake throughout the study duration. Data collected from the application will be the primary measure of adherence to dietary changes.
  Arms: Calorie Restriction - Communication Standard of Care; Calorie Restriction - Frequent Patient Communication

SUMMARY:
This is a pragmatic, single-blinded randomized trial of improving adherence to dietary interventions in patients with MS who are receiving monthly natalizumab infusions.

DETAILED DESCRIPTION:
MS affects at least 400,000 people in the US alone, and its incidence has increased in the past 50 years, likely due to changing environmental risk factors. Recent research suggests that diet may be a critical factor in the development of MS. The "Western diet", high in sugar, fat, and salt, may influence MS risk and progression by directly affecting the immune system, altering gut bacteria, and changing metabolism.

Studying patients with MS who are overweight and obese may be relevant as obesity can cause chronic low-grade inflammation, potentially worsening MS symptoms. Diet modification represents an interesting potential therapy for MS, particularly calorie restriction and fasting, which have been associated with reduced markers of inflammation. In addition to these direct effects, weight optimization may lead to improvements in MS-related symptoms, like fatigue, and overall quality of life.

This is a single-blinded randomized trial of adherence to a dietary intervention in patients with MS who are receiving monthly natalizumab infusions. The study will evaluate how use of technology may help patients with MS adhere to a calorie restricted diet. It will also evaluate the effect of weight loss on fatigue and quality of life in patients with MS. A second part of the study will evaluate if shortening the period during the day in which people consume their typical food amounts leads to improvements in patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 25 kg/m^2 for calorie restriction study
* BMI < 25 kg/m^2, or ≥ 25 kg/m^2 if participant was unwilling to enroll in calorie restriction study
* Smartphone with the ability to download and use the LoseIt! application (calorie restriction only)
* Smartphone with the ability to take and store photos (calorie timing only)

Exclusion Criteria:

* History of diabetes requiring medication
* Currently pregnant or breastfeeding
* History of an eating disorder
* Currently taking warfarin
* History of major surgery within past 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mowry, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No
Individual participant's data will not be shared

REFERENCES:
- [Derived] Roman SN, Fitzgerald KC, Beier M, Mowry EM. Safety and feasibility of various fasting-mimicking diets among people with multiple sclerosis. Mult Scler Relat Disord. 2020 Jul;42:102149. doi: 10.1016/j.msard.2020.102149. Epub 2020 May 6. PMID 32408153

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Timing Restriction | No Diet Change
Started | 15 | 12 | 14 | 13
Baseline Study Visit | 10 | 9 | 14 | 12
3 Month Study Visit | 7 | 8 | 12 | 11
Completed | 7 | 8 | 12 | 11
Not Completed | 8 | 4 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 2 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Calorie Restriction - Frequent Patient Communication: Participants select to restrict calories continuously (25% daily) or intermittently (76% twice per week) for the 6-month study period. Weekly informational and supportive text messages will be sent to patients, encouraging adherence to the calorie restriction diet.
- Calorie Restriction - Communication Standard of Care: Participants select to restrict calories continuously (25% daily) or intermittently (76% twice per week) for the 6-month study period. Participants will not receive additional support or interaction from the study team apart from the scheduled study visits.
- Timing Restriction: Patients who do not qualify for, or do not wish to complete, the calorie restriction diet, may be randomized to time restriction. In this arm, participants restrict their calorie intake to an 8-hour interval each day, providing time for a 16-hour fast between intervals.
- No Diet Change: Patients who do not qualify for, or do not wish to complete, the calorie restriction diet, may be randomized to not make any diet changes. This group is instructed to continue eating their normal diet throughout the 6-month study period.
- Total: Total of all reporting groups
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Timing Restriction | No Diet Change | Total
Number analyzed (Participants) | 10 | 9 | 12 | 12 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.10 (6.00) | 31.18 (3.79) | 39.83 (10.94) | 43.42 (11.77) | 41.73 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 10 | 10 | 37
  Male | 0 | 2 | 2 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 7 | 8 | 7 | 28
  African American | 3 | 0 | 4 | 4 | 11
  Non-White Hispanic | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 0 | 1
  Other | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 12 | 12 | 43
Weight [Mean (Standard Deviation); unit: kg] | 92.58 (17.26) | 82.76 (16.89) | 66.25 (8.12) | 70.13 (16.06) | 76.91 (17.73)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.04 (6.52) | 30.22 (4.78) | 24.28 (3.16) | 25.86 (6.22) | 28.00 (6.21)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 110.22 (19.31) | 102.16 (13.05) | 87.58 (11.63) | 89.38 (12.58) | 96.4 (16.68)
Hip Circumference [Mean (Standard Deviation); unit: cm] | 118.36 (14.85) | 109.80 (7.15) | 99.08 (7.24) | 100.26 (11.01) | 106.14 (12.84)
Patient-Determined Disability Score [Mean (Standard Deviation); unit: scores on a scale] — The Patient-Determine Disability Scale (PDDS) measures level of disability from multiple sclerosis as reported by the patient. The scale ranges from a minimum of 0 (No disability - "I may have some mild symptoms, mostly sensory due to MS, but they do not limit my activity") to a maximum of 8 (Bedridden - "Unable to sit in a wheelchair for more than one hour"). Lower values on this scale indicate less disability from multiple sclerosis. A reduction in PDDS over the study period indicates a better outcome, or improvement in disability/symptoms from MS, among participants.
  scores on a scale | 1.09 (1.62) | 1.89 (1.54) | 2.58 (1.56) | 3.00 (2.14) | 2.21 (1.82)
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue-MS Score [Mean (Standard Deviation); unit: scores on a scale] — The Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue is a 95-item question bank to evaluate fatigue in a variety of chronic conditions. The PROMIS-FatigueMS is a subset of 8 questions from the question bank, which have been validated to measure fatigue specifically in people with multiple sclerosis. Individual items are scored on a 5-point Likert scale, and the total score is the sum of individual items, with a minimum score of 8 and maximum score of 40. Lower scores indicate less fatigue; reduction in score over 6 months indicates a better outcome.
  scores on a scale | 21.40 (9.30) | 22.94 (7.67) | 22.50 (6.49) | 20.96 (9.46) | 21.91 (8.05)
Pittsburgh Sleep Quality Index Score [Mean (Standard Deviation); unit: scores on a scale] — The Pittsburgh Sleep Quality Index (PSQI) is an instrument used to measure the quality and sleeping pattern of adults. It differentiates "poor" from "good" sleep quality, and the total score is calculated from the sum of seven components, each scored from 0 to 3. The minimum total score is 0 and the maximum total score is 21. A total score equal to or greater than 5 units indicates "poor" quality sleep, while a score of 0-4 indicates "good" quality sleep; lower scores indicate better sleep quality.
  scores on a scale | 8.50 (4.56) | 6.56 (4.22) | 7.75 (5.96) | 8.17 (4.76) | 7.79 (4.74)
Quality of Life [Mean (Standard Deviation); unit: scores on a scale] — The Functional Assessment in Multiple Sclerosis (FAMS) is an instrument that measures quality of life among people with MS. It contains 44 questions scored on a 5-point Likert scale in 6 areas: mobility, symptoms, emotional wellbeing, general contentment, thinking/fatigue, and family/social wellbeing. Subscores are the sum of responses in that section, and the total FAMS score is the sum of all subscores. Minimum total score is 0 and maximum total score is 176, where a higher score indicates better quality of life. Increase in score over the study period indicates a better outcome.
  scores on a scale | 174.73 (38.05) | 162.49 (34.24) | 145.81 (36.48) | 144.86 (49.44) | 156.02 (40.72)
Rosenberg Self-Esteem Score [Mean (Standard Deviation); unit: scores on a scale] — The Rosenberg Self-Esteem Scale (RSES) is a 10-item scale that measures global self-worth using a 4-point Likert scale to ask about negative and positive feelings about the self. Individual items are summed to calculate the total score. Minimum score is 0 and maximum score is 30. Higher scores indicate higher/better self-esteem. Scores between 15 and 25 are considered within the normal range, while scores below 15 indicates poor self-esteem. An increase in RSES score over 6 months indicates a better outcome, or improved self-esteem, among participants.
  scores on a scale | 21.65 (7.89) | 25.11 (2.42) | 24.33 (1.56) | 24.17 (2.69) | 23.83 (4.31)

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Number of participants adhering to the prescribed dietary intervention at the end of the 6-month study period.
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Timing Restriction | No Diet Change
Number analyzed (Participants) | 10 | 9 | 12 | 12
Participants | 2 | 6 | 10 | 12

2. Secondary Outcome: Body Mass Index (BMI)
Description: Change in body mass index from baseline to 6 months.
Time Frame: Baseline and 6 months
Population: 5 out of the initial 43 participants dropped out of the study voluntarily
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Calorie Restriction - Frequent Patient Communication: Participants selected to restrict calories continuously (25% daily) or intermittently (76% twice per week) for the 6-month study period. Weekly informational and supportive text messages was sent to patients, encouraging adherence to the calorie restriction diet.
- Calorie Restriction - Communication Standard of Care: Participants selected to restrict calories continuously (25% daily) or intermittently (76% twice per week) for the 6-month study period. Participants did not receive additional support or interaction from the study team apart from the scheduled study visits.
- Time Restriction: Participants adhering to a daily 16-hour fasting period, so they restrict all calorie intake to an 8-hour interval each day.
- No Diet Change: Participants make no changes to their normal diet.
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Time Restriction | No Diet Change
Number analyzed (Participants) | 7 | 8 | 12 | 11
kg/m^2 | -0.83 (1.77) | -1.03 (1.13) | 0.04 (1.09) | -0.22 (0.70)

3. Secondary Outcome: Weight Change
Description: Change in participant weight over the 6-month study period
Time Frame: Baseline and 6 months
Population: 5 out of the initial 43 participants dropped out of the study voluntarily
Measure: Mean (Standard Deviation); unit: KG
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Time Restriction | No Diet Change
Number analyzed (Participants) | 7 | 8 | 12 | 11
KG | -2.15 (4.72) | -2.85 (3.06) | 0.12 (3.02) | -0.52 (1.88)

4. Secondary Outcome: Weight Change Among Adherent Participants
Description: The change in weight over 6 months among participants were remained adherence to the calorie restriction diet versus those who admitted to non-compliance by the end of the study period.
Time Frame: Baseline and 6 months
Population: Discrepancy in numbers is due to non-completers. 5 out of the initial 43 participants dropped out of the study voluntarily
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Calorie Restriction - Adherent Participants: Participants still following a calorie restriction diet, continuous or intermittent, at the end of the 6 month period. Includes participants in both randomization arms (frequent communication and standard of care).
- Calorie Restriction - Non-Adherent Participants: Participants who started in either the frequent communication or communication standard of care arms, following a calorie restriction diet, but who stopped the diet prior to the end of the 6-month study period.
Arm/Group | Calorie Restriction - Adherent Participants | Calorie Restriction - Non-Adherent Participants
Number analyzed (Participants) | 8 | 8
kg | -4.97 (4.06) | -0.22 (2.38)

5. Secondary Outcome: Functional Assessment in MS Score
Description: The Functional Assessment in Multiple Sclerosis (FAMS) is an instrument that measures quality of life among people with MS. The instrument contains 44 questions scored on a 5-point Likert scale in 6 areas: mobility, symptoms, emotional wellbeing, general contentment, thanking/fatigue, and family/social wellbeing. Subscores for each area is calculated as the sum of responses in that section, and the total FAMS score is the sum of all subscores. Minimum total score is 0 and maximum total score is 176, where a higher score indicates better quality of life. Increase in the FAMS score over the study period indicates a better outcome, or improved quality of life, among participants.
Time Frame: Baseline and 6 months
Population: 5 out of the initial 43 participants dropped out of the study voluntarily
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Time Restriction | No Diet Change
Number analyzed (Participants) | 8 | 7 | 12 | 11
scores on a scale | -3.96 (28.38) | 5.73 (18.62) | 5.42 (21.71) | 2.17 (23.90)

6. Secondary Outcome: Fatigue
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue is a question bank of 95 items validated to evaluated fatigue in a variety of chronic conditions. The PROMIS-FatigueMS is a subset of 8 questions from the question bank, which have been validated to measure fatigue in people with multiple sclerosis. Individual items are scored on a 5-point Likert scale, and the total score is the sum of individual items, with a minimum score of 8 and maximum score of 40. Lower scores indicate less fatigue, while higher scores indicate more fatigue. Reduction in score over 6 months indicates a better outcome, or improved fatigue among participants.
Time Frame: Baseline and 6 months
Population: Discrepancy in numbers is due to non-completers
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Time Restriction | No Diet Change
Number analyzed (Participants) | 7 | 8 | 12 | 11
scores on a scale | -3.38 (3.96) | -2.07 (4.60) | -0.58 (5.35) | 1.18 (5.42)

7. Secondary Outcome: Sleep Quality
Description: The Pittsburgh Sleep Quality Index (PSQI) is an instrument used to measure the quality and sleeping pattern of adults. It differentiates "poor" from "good" sleep quality, and the total score is calculated from the sum of seven components, each scored from 0 to 3. The minimum total score is 0 and the maximum total score is 21. A total score equal to or greater than 5 units indicates "poor" quality sleep, while a score of 0-4 indicates "good" quality sleep; lower scores indicate better sleep quality. Decrease in PSQI score indicates a better outcome, or improved sleep quality, among study participants.
Time Frame: Baseline and 6 months
Population: 5 out of the initial 43 participants dropped out of the study voluntarily
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Time Restriction | No Diet Change
Number analyzed (Participants) | 7 | 8 | 12 | 11
scores on a scale | -1.33 (3.08) | -0.75 (2.19) | -1.50 (3.78) | -0.73 (3.95)

8. Secondary Outcome: Self-esteem
Description: The Rosenberg Self-Esteem Scale (RSES) is a 10-item scale that measures global self-worth using a 4-point Likert scale to ask about negative and positive feelings about the self. Individual items are summed to calculate the total score. Minimum score is 0 and maximum score is 30. Scores between 15 and 25 are considered within the normal range, while scores below 15 indicates poor self-esteem. An increase in RSES score over 6 months indicates a better outcome, or improved self-esteem, among participants.
Time Frame: Baseline and 6 months
Population: 5 out of the initial 43 participants dropped out of the study voluntarily
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Time Restriction | No Diet Change
Number analyzed (Participants) | 7 | 8 | 12 | 11
scores on a scale | 0.39 (2.06) | -1.00 (1.93) | -1.00 (2.70) | 1.41 (3.53)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through the duration of the 6-month intervention period for each participant. Including all participants, this data was collected from October 2016 until the end of June 2017.
Arm/Group | Calorie Restriction - Frequent Patient Communication | Calorie Restriction - Communication Standard of Care | Timing Restriction | No Diet Change
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/10 | 0/9 | 0/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calorie Restriction - Frequent Patient Communication (N=10) | Calorie Restriction - Communication Standard of Care (N=9) | Timing Restriction (N=12) | No Diet Change (N=12)
Migraine (Nervous system disorders) | 1 (1) | 0 | 0 | 0 — One patient with a known history of migraine headaches experienced migraines on fasting days for the intermittent calorie restriction option, and self-discontinued the dietary intervention.

LIMITATIONS AND CAVEATS:
Limited sample size; Participants were enrolled from one treatment center, limited to patients with relapsing-remitting subtype of MS on natalizumab treatments; Calorie and timing data were self-reported by participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT02846558/Prot_SAP_000.pdf